CLINICAL TRIAL: NCT00754832
Title: A Double-blinded, Placebo-controlled Crossover Pilot Study of American Ginseng Treatment for Multiple Sclerosis Related Fatigue
Brief Title: American Ginseng Treatment for Multiple Sclerosis Related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Ruth Whitham, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1357
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; fatigue; ginseng
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Period 1 with Ginseng therapy intervention; Washout Period with no drug; Period 2 with placebo
  Interventions: Drug: American ginseng extract HT-1001; Drug: placebo
- 2 (Experimental): Period 1 with placebo; Washout period with no drug; Period 2 with ginseng therapy intervention
  Interventions: Drug: American ginseng extract HT-1001; Drug: placebo

INTERVENTIONS:
Drug: American ginseng extract HT-1001 — Ginseng HT-1001 was dosed at 100 mg orally per day initially, increased after one week to 200 mg per day, then further increased the next week to 400 mg per day as tolerated. Subjects were then maintained on 400 mg per day or the maximum tolerated dose for the remainder of the 6 week treatment period.
Drug: placebo — Placebo capsules were identical to the study drug and were dose escalated to match the study drug. Subjects were maintained on placebo capsules for the remainder of the 6 week treatment period.
  Other Names: placebo (matched capsules to ginseng drug)

SUMMARY:
This research project will determine the safety and tolerability of ginseng in subjects with MS and will gather preliminary data on the efficacy of ginseng vs placebo for the treatment of MS fatigue.

DETAILED DESCRIPTION:
Fatigue is a major cause of disability in MS and is associated with a reduced quality of life. Treatment options for MS fatigue include central nervous system stimulants and amantadine. These medications are of limited efficacy, are often poorly tolerated, and can be expensive. Ginseng may represent a novel approach to treating MS fatigue. Ginseng has been tested in clinical trials for its ability to improve mental alertness and fatigue. However, there have been no published clinical trials addressing the effects of ginseng in subjects with MS, even though many people with MS use ginseng and report deriving benefit from it.

This double-blinded, placebo controlled crossover pilot study will determine the safety and tolerability of ginseng in subjects with MS and will gather preliminary data on the efficacy of ginseng vs. placebo for the treatment of MS fatigue. Additionally, the project will collect information on the impact of ginseng on cognition, stress, actigraphy, salivary cortisol, differential cytokine response, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* MS as diagnosed by the McDonald criteria
* Complaint of fatigue that has been persistent for at least 2 months
* FSS score of 4 or greater;
* Age 18-70.

Exclusion Criteria:

* Use of ginseng or stimulants in the prior 6 weeks
* Acute treatment with glucocorticoids in the prior 6 weeks
* BDI >31
* Significant MS exacerbation in prior 30 days
* Diabetes
* Uncontrolled hypertension
* Other serious medical disease, pregnancy or breastfeeding
* Breast disease
* Abnormal bleeding or clotting disorder
* Current use of warfarin, albendazole, nifedipine, digoxin, bumetadine, selegiline, isocarboxazid, or phenelzine
* Current use of lasix for poorly controlled hypertension or congestive heart failure
* Current drug or alcohol abuse; inability to complete the self report forms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-09; Primary Completion 2008-09 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Whitham, M.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Kim E, Cameron M, Lovera J, Schaben L, Bourdette D, Whitham R. American ginseng does not improve fatigue in multiple sclerosis: a single center randomized double-blind placebo-controlled crossover pilot study. Mult Scler. 2011 Dec;17(12):1523-6. doi: 10.1177/1352458511412062. Epub 2011 Jul 29. PMID 21803872
- [Derived] Kim E, Lovera J, Schaben L, Melara J, Bourdette D, Whitham R. Novel method for measurement of fatigue in multiple sclerosis: Real-Time Digital Fatigue Score. J Rehabil Res Dev. 2010;47(5):477-84. doi: 10.1682/jrrd.2009.09.0151. PMID 20803391

RESULTS

PARTICIPANT FLOW:
Groups:
- Ginseng First Then Placebo: ginseng 100 mg daily escalating to 400 mg daily for 6 weeks followed by 2 weeks washout, then placebo 1 cap daily escalating to 4 caps daily for 6 weeks
- Placebo First Then Ginseng: placebo 1 cap daily escalating to 4 caps daily for 6 weeks followed by 2 weeks washout, then ginseng 100 mg daily escalating to 400 mg daily for 6 weeks
Period: First 6 Weeks Intervention
Arm/Group | Ginseng First Then Placebo | Placebo First Then Ginseng
Started | 26 | 30
Completed | 18 | 28
Not Completed | 8 | 2
Period: 2 Weeks Washout
Arm/Group | Ginseng First Then Placebo | Placebo First Then Ginseng
Started | 18 | 28
Completed | 17 | 26
Not Completed | 1 | 2
Period: Second 6 Weeks Intervention
Arm/Group | Ginseng First Then Placebo | Placebo First Then Ginseng
Started | 17 | 26
Completed | 17 | 24
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intent to Treat Study Population: all participants who received at least one dose of either placebo or ginseng in this crossover trial
Arm/Group | Intent to Treat Study Population
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.5 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Severity Scale
Description: The Fatigue Severity Scale (FSS)is a self-administered instrument that includes 9 items rated on a 7-point scale, measuring fatigue severity. The subject is asked to score each statement, based on how the statement applied to them over the preceding week. The fatigue severity score is the average of the scores on the 9 questions; scores range from 1-7, with lower scores indicating less fatigue.
Time Frame: after 6 weeks of intervention
Population: intention to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Ginseng: ginseng 100 mg daily escalating to 400 mg daily for 6 weeks
- Placebo: placebo 1 tab daily escalating to 4 tabs daily for 6 weeks
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 47 | 47
units on a scale | 5.5 (1.3) | 5.5 (1.3)

2. Secondary Outcome: Modified Fatigue Impact Scale
Description: 21 item scale, score range 0-84, lower scores indicate less fatigue
Time Frame: 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 47 | 47
units on a scale | 42.7 (15.7) | 43.7 (16.7)

3. Secondary Outcome: Realtime Digital Fatigue Score
Description: fatigue scored on 0-10 scale with higher scores indicating more fatigue
Time Frame: 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginseng | Placebo
Number analyzed (Participants) | 47 | 47
units on a scale | 4.2 (1.6) | 4.2 (1.8)

ADVERSE EVENTS:
Arm/Group | Ginseng | Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 5/56 | 4/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ginseng (N=56) | Placebo (N=56)
rash (Skin and subcutaneous tissue disorders) | 3 | 0
insomnia (Psychiatric disorders) | 3 | 4
headache (Nervous system disorders) | 3 | 1
nausea (Gastrointestinal disorders) | 4 | 4
flu like syndrome (General disorders) | 3 | 2
upper respiratory infection (Infections and infestations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes